CLINICAL TRIAL: NCT01268228
Title: COronary SIde Branch Residual IschemiA and COllateralization Assessment Study (COSIBRIA & Co Study)
Brief Title: Intracoronary Electrocardiogram (ECG) and Myonecrosis After Bifurcation Stenting
Acronym: COSIBRIA&CO
Status: Completed | Type: Observational
Sponsor: University National Heart Hospital (Other)
Responsible Party: Principal Investigator, Dobrin Vassilev, Dobrin Vassilev MD, PhD, University National Heart Hospital
Other Study IDs: ICECG-12-2010
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Periprocedural Myonecrosis
Keywords: intracoronary ECG; coronary bifurcation stenosis; side branch compromise; Periprocedural myonecrosis during coronary bifurcation lesion stenting assessed with ic ECG

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Residual ic ECG ST elevation in SB
- Residual ic ECG ST elevation in MB

SUMMARY:
The coronary bifurcation lesions pose a therapeutic problem with high rates of periprocedural complications, higher rates of in-stent restenosis and stent thrombosis. These are lesions where stenting is not superior in comparison to balloon angioplasty in regard to side branch. It was demonstrated many times, in literature and in daily practice, that angiographically high grade ostial side branch stenosis is not flow limiting and do not cause ischemia, therefore do not require treatment. From the other side, our own data with MRI before and after bifurcation PCI demonstrated that occurrence of angiographic stenosis more than 70% in diameter is associated with periprocedural myonecrosis in the region of side branch. This fact puts a very important question about the mechanisms of this myonecrosis. If the jailed side branch has no significant flow limiting stenosis, but there is some degree of residual ischemia, which after some period of persistence could lead to myonecrosis, will mean that more aggressive treatment of ostial stenosis is needed. It is interesting that the strategy of treatment is very important, because techniques with second stent implantation (with primary purpose to limit SB ischemia) are associated with higher grade of troponin increase. Of course this is association and not causality, despite that in randomized study (NORDIC I) it was confirmed also.

It is without explanation the fact of rare occurrence of significant (flow limiting, FFR <.75) stenosis appearance (less than 40% in side branches with ostial stenosis more than 75%) and almost 50% periprocedural myonecrosis detected in the side branch areas. One working hypothesis is that stent implantation and related episode of ischemia induces prolonged vasospasm, resulting in prolonged ischemia. Thus, the ostial stenosis could be non-significant as estimated and registered by FFR, but on microcirculatory lever ischemia could persist is small areas for which available flow is not sufficient despite that global regional flow is deemed sufficient. It is also possible that those patients have not enough recruitable collaterals. It is also possible that both factors act together.

Although FFR is useful for assessing the degree of ischemia caused by a coronary lesion, it cannot give information as to whether this ischemia may be clinically significant or not, i.e. whether the ischemia affects a large territory. Therefore, it can be implicated that FFR may not be useful in predicting clinically meaningful ischemia in a specific side branch vessel.

The intracoronary electrocardiography (i.c. ECG) is a very sensitive method for ischemia detection. The i.c. ECG reacts earlier on ischemia; the changes are much more prominent and easy to register. The wire tip could be positioned directly in different regions and thus to "map" regional ischemia. In most of the studies and from our own observations became evident that when surface ECG do not react the i.c. ECG demonstrates significant changes in ST-segment and QRS complex. Moreover, the registration of i.c. ECG is very cheap and needs only an adapter connecting coronary wire end and ECG. An i.c. ECG also can differentiate residual ischemic changes in distal main vessel and side branch as sources of prolonged ischemia, respectively - source of periprocedural myonecrosis.

The objective of this study is to evaluate the clinical significance of side branch vessel by occluding the blood flow with a 1-minute balloon occlusion. We will also assess whether there is any change in ECG (i.c. and 12-lead surface records) on balloon occlusion and relation with periprocedural myonecrosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject at least 18 years of age.
* Subject able to verbally confirm understandings of risks, benefits of receiving PCI for true bifurcation lesions, and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
* Target main branch lesion(s) located in a native coronary artery with diameter of ≥ 2.5 mm and ≤ 4.5 mm. Target side branch lesion(s) located in a native coronary artery with diameter of ≥ 2.0 mm.
* Target lesion(s) amenable for PCI with balloon angioplasty of the side branch.

Exclusion Criteria:

* Subjects with significant ST-T change (≥ 1mm).
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* Subjects who refuse to give informed consent.
* Subjects with the following angiographic characteristics: left main coronary artery stenosis, total occlusion before occurrence of SB, lesion of interest located at infarct-related artery.
* Subjects with LVEF < 30%.
* Subjects with moderate or severe degree valvular heart disease or primary cardiomyopathy.
* LBBB, RBBB, atrial fibrillation/flutter with no identifiable isoelectric line.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Significant, >50% diameter stenosis artery scheduled for stent insertion at the main vessel (Medina types: 1xx, x1x, 11x);
  * Side branch vessel at least 2.0mm
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2011-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
periprocedural myonecrosis | 48 hours
  Periprocedural myonecrosis - > ULN, 3-5 ULN, >5x ULN; measure - Trponin I & CK-MB

SECONDARY OUTCOMES:
Major cardiovascular events: death, MI, TLR | 12 months
TLR - target lesion revascularization | 12 months
  The rate of repeated PCI procedures obeing stent + 5mm territory from stent edges during follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Dobrin Vassilev, MD, PhD, Principal Investigator — University National Heart Hospital
Locations (3):
- Bulgaria (2):
  - Medica Core Heart Hopsital, Rousse, Bulgaria
  - University National Heart Hospital, Sofia
- Central Hospital of the Internal Affairs and Administration Ministry, Warsaw, Poland, Poland